CLINICAL TRIAL: NCT00802022
Title: Effect of Spinal Cord Stimulation in Painful Diabetic Polyneuropathy (PDP Study) A Pilot Study
Brief Title: Effect of Spinal Cord Stimulation in Painful Diabetic Polyneuropathy
Acronym: SCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Prof. dr. M. van Kleef, Maastricht University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEC 08-2-118
Record Dates: First submitted 2008-12-03; First posted 2008-12-04 (Estimated); Last update posted 2010-07-08 (Estimated); Status verified 2010-07

CONDITIONS: Diabetic Neuropathies
Keywords: diabetic neuropathies; electric stimulation therapy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: spinal cord stimulation — The intervention is spinal cord stimulation and will be used for 2 weeks trial stimulation. After clinical successful pain relief (50% of more pain reduction)a definite spinal cord system will be implanted.
  Other Names: Medtronic leads and neurostimulator (CE mark 0123)

SUMMARY:
Rationale: Diabetic neuropathy is one of the most common complications of Diabetes Mellitis (DM). Pain is a common symptom of diabetic neuropathy, affecting 11-34% of patients suffering form DM. The current available medication often provides insufficient pain relief and/or has unacceptable side effects. Spinal cord stimulation (SCS) has been used for over 30 years to treat neuropathic pain. Various small clinical studies have shown a beneficial effect of SCS on pain in PDP.

Objective: This study is a preparation to a RCT to investigate whether SCS is a good indication in patients which suffer from pain with moderate-to-severe PDP in the lower limbs. The main objective of this study is whether SCS leads to sufficient pain relief and to obtain insight into the working mechanism of SCS. The hypothesis is that the effect SCS is most effective in patients without major sensory deficits. Furthermore, practical feasibility of the test procedures described in the study protocol will be examined, including the questionnaires to be filled out by the patient. Also, technical feasibility of SCS will be investigated. Besides the feasibility, the possibility of predicting successful pain relief by SCS by classifying patients according to the Michigan Diabetic Neuropathy Score will be assessed. Furthermore, possible other predictors for successful pain relief by SCS will be defined. Study design: the study is a pilot study in preparation to a RCT to investigate the effect of spinal cord stimulation on pain in moderate-to-severe PDP patients.

Study population: patients suffering from moderate-to-severe PDP in the lower limbs as diagnosed by clinical symptoms and supported by the Michigan Diabetic Neuropathy Score.

Intervention: patients will receive 2 weeks of trial stimulation and best (drug) treatment as usual.

Main study parameters/endpoints: Main study parameter is the pain score as measured by a numeric rating scale (NRS) according to Jensen and a Patient Global Impression of Change for pain measured on a 7-point Likert scale.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: SCS related risks include: lead migration (14%), lead breakage (7%), implanted pulse generator migration (1%), loss of therapeutic effect, lost or unpleasant paresthesias (12%), infection or wound breakdown (10%), Pain at IPG incision site (12%), IPG pocket fluid collection (5%).

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe PDP in the lower limbs

  * The pain intended to treat has been present for more than 12 months
  * Previous treatment has been unsuccessful (insufficient pain relief and/or unacceptable side-effects) with drugs from the following drug categories:
  * Amitriptyline or an other tricyclic antidepressant and/or
  * Pregabalin (Lyrica), Gabapentin (Neurontin) or Carbamazepine and/or
  * Duloxetine (Cymbalta) and/or
  * Tramadol or strong opioids Patients were treated with 3 drugs from the above mentioned drug categories and followed the treatment algorithm for painful diabetic polyneuropathy according to Jensen. Each drug is tried for 3 weeks and dose is raised once. By insufficient pain relief and/or unacceptable side-effects, the drug treatment was stopped. Patients reached a steady state in medication use and it is not allowed to change the use of medication during the study.
* Mean pain intensity should be 5 or higher measured on a numeric rating scale (NRS), which will be scored 3 times per day during 4 days according to Jensen.
* Patients age is between 18 and 75 years.

Exclusion Criteria:

* The patient has had neuromodulation therapy during the month before the intake
* The patient has ever had neuromodulation
* Neuropathic pain prevalent in the upper limbs (NRS above 3)
* Neuropathy or chronic pain of other origin than diabetes mellitus (NRS above 3)
* Addiction: drugs, alcohol (5E/day) and/or medication

  * Drugs: cocaine, heroine, marihuana,
  * Alcohol: wine, beer, liquor.
  * Medication: benzodiazepines, morphine receptor agonists.
* Insufficient cooperation from the patient (little motivation, understanding or communication)
* Blood clotting disorder
* Immune deficiency (HIV-positive, corticosteroids with a dose equivalent to prednisolone 10 mg, immunosuppressive, etc.)
* Peripheral vascular disease, no palpable peripheral pulsations at the feet (inclusion is possible if pulsations are absent, but ankle/brachial index is between 0.7 and 1.2 in both feet)
* Active foot ulceration
* Life expectancy shorter than 1 year
* Pacemaker
* Local infection or other skin disorders at site of incision
* Psychiatric disorders
* Pregnancy
* Severe cardiac or pulmonary failure (NYHA classification II or higher)
* Unstable blood glucose control (change in HbA1c more than 1,0% (absolute value) in three months prior to inclusion)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-01; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Pain intensity measured on a weighted NRS according to Jensen and a PGIC for pain measured on a 7-point Likert scale. | Baseline, 2 weeks after trial stimulation, 3, 6 and 12 months

SECONDARY OUTCOMES:
The practical- and technical feasibility of the procedures, predicting successful pain relief by SCS by classifying patients according to the MDNS. Define possible other predictors for successful pain relief. | Baseline, 2 weeks after trial stimulation, 3, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maarten van Kleef, prof. dr., Principal Investigator — Maastricht University Hospital
Locations (1):
- Maastricht University Hospital, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Tesfaye S, Watt J, Benbow SJ, Pang KA, Miles J, MacFarlane IA. Electrical spinal-cord stimulation for painful diabetic peripheral neuropathy. Lancet. 1996 Dec 21-28;348(9043):1698-701. doi: 10.1016/S0140-6736(96)02467-1. PMID 8973433
- [Background] de Vos CC, Rajan V, Steenbergen W, van der Aa HE, Buschman HP. Effect and safety of spinal cord stimulation for treatment of chronic pain caused by diabetic neuropathy. J Diabetes Complications. 2009 Jan-Feb;23(1):40-5. doi: 10.1016/j.jdiacomp.2007.08.002. Epub 2008 Apr 16. PMID 18413161
- [Derived] van Beek M, Geurts JW, Slangen R, Schaper NC, Faber CG, Joosten EA, Dirksen CD, van Dongen RT, van Kuijk SMJ, van Kleef M. Severity of Neuropathy Is Associated With Long-term Spinal Cord Stimulation Outcome in Painful Diabetic Peripheral Neuropathy: Five-Year Follow-up of a Prospective Two-Center Clinical Trial. Diabetes Care. 2018 Jan;41(1):32-38. doi: 10.2337/dc17-0983. Epub 2017 Nov 6. PMID 29109298